CLINICAL TRIAL: NCT05880641
Title: No-profit, Pilot, Observational, Multicentric, Prospective Study on the Use of Shockwave M5+ IVL Catheter (Intravascular Lithotripsy) in Hostile and Calcified Iliac Access to Facilitate Aortic Endovascular Repair. SHOCK-ACCESS STUDY.
Brief Title: Use of Shockwave M5+ IVL Catheter (Intravascular Lithotripsy) in Hostile and Calcified Iliac Access
Acronym: SHOCK-ACCESS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: EndoCore Lab s.r.l. (Other)
Collaborators: Fondazione Italiana Vascolare (Other)
Responsible Party: Sponsor
Other Study IDs: IVL 022022
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Aortic Diseases; Aorto-Iliac Atherosclerosis; Peripheral Arterial Disease
Keywords: Aortic Disease; Intravascular Lithotripsy; Hostile Access
MeSH Terms: conditions — Aortic Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will evaluate, in a controlled setting, the efficacy and safety of the intravascular lithotripsy using Shockwave™ M5+ Peripheral Intravascular Lithotripsy Catheter to facilitate delivery of aortic large-bore devices in iliac calcified access.

DETAILED DESCRIPTION:
This study is designed as no-profit, pilot, observational, multicentric, prospective study.

All eligible subjects for undergoing intervention with Shockwave™ M5+ Peripheral Intravascular Lithotripsy Catheter (IVL) at sites participating in the study will be considered for enrolment and will be asked to give consent prior to participating.

Subjects will be considered enrolled in the study at the time written informed consent is given to the use of their personal data. Once patients are enrolled, their demographics, medical history, disease-relevant conditions, treatment details and outcomes will be collected for up to 12 months from the procedure.

The study will collect information about the medical care patients receive during their planned procedure. No additional testing or procedures will be done.

The procedure with Shockwave™ M5+ Peripheral Intravascular Lithotripsy Catheter (IVL) will be performed as per the current instructions for use.

After discharge all patients will attend clinic visits at 30 days (±14 days), 6 months (±30 days),12 months (±30 days).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Patient (or their legal representative) understands the nature of the procedure and provides written informed consent, prior to enrolment in the study;
* Patient presenting with aortic disease indicated for endovascular treatment considered unfeasible based on severely calcified iliac access and outer diameter of the "ideal" aortic endograft at onset of the procedure (considering the main body and/or contralateral limb in case of iliac distal landing zone);
* Patients presenting a ratio > 0.2 between outer diameter of the aortic stent graft delivery system (OD-SG) and minimum lumen diameter (MLD); decision concerning SG will be taken balancing the lower profile on the market and the better graft fit for patient's anatomy;
* Patients presenting calcium grade 3 or 4 accordingly to 360° coronary classification (grade 1 = 0-90°, grade 2 = 90°-180°; grade 3 = 180°-270°; grade 4 = 270°-360°);
* Patients presenting a lesion length > 20 mm, intended as the sum of all calcified iliac lesions between two endpoints, from the aortic bifurcation up to the proximal common femoral artery (CFA);
* Patients eligible for treatment with Shockwave M5+ IVL device;
* Patients presenting with aortic disease indicated for endovascular treatment associated or not to aorto-iliac occlusive disease (Rutherford classification score II - VI for chronic limb ischemia);
* Patients compliant with the conduct of follow-up visits according to the timelines specified in the protocol.

Exclusion Criteria:

* Bilateral Iliac Occlusion;
* Urgent setting with presence of iliac thrombus (acute limb ischemia);
* Any patient considered to be hemodynamically unstable at procedure onset;
* Patients refusing treatment;
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated;
* Patients with a history of prior life-threatening contrast medium reaction;
* Life expectancy of less than twelve months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aortic diseases (abdominal, thoracic or thoraco-abdominal, aneurysms, dissections, PAU, IMH) with hostile iliac access (calcified and narrowed) associated or not to aorto-iliac occlusive disease (AIOD).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Minimum Lumen Diameter (MLD) Gain | Baseline, Day 1
  Minimum Lumen Diameter (MLD) Gain defined as the difference between MLD post-procedure and MLD pre-procedure.

SECONDARY OUTCOMES:
Technical success of Shockwave™ M5+ IVL | Day 1
  Technical success of Shockwave™ M5+ IVL defined as the successful delivery and positioning of the aortic endograft;
Composite of Freedom from iliac complications | Day 1, 1 Month
  Freedom from iliac complications composite (flow-limiting dissections, distal embolizations, trauma, rupture) at day 1, 30 days
Freedom from vessel flow-limiting dissections | Day 1, 1 Month
  Freedom from vessel flow-limiting dissections at day 1 and 1 Month
Freedom from vessel distal embolization | Day 1, 1 Month
  Freedom from vessel distal embolization at day 1 and 1 Month
Freedom from vessel trauma | Day 1, 1 Month
  Freedom from vessel trauma at day 1 and 1 Month
Freedom from vessel rupture | Day 1, 1 Month
  Freedom from vessel rupture at day 1 and 1 Month
Freedom from bailout manoeuvres | Day 1
  Freedom from bailout manoeuvres (stenting/endoconduits) at day 1
Freedom from iliac secondary procedures | Day 1
  Freedom from iliac secondary procedures other than IVL at day 1
Freedom from access-site adjunctive/secondary procedures; | Day 1
  Freedom from access-site adjunctive/secondary procedures
Primary patency of the target lesion for each iliac axis treated with IVL | 1 month, 6 months, 12 months
  Primary patency of the target lesion for each iliac axis treated with IVL: defined as a lesion without a severe restenosis/occlusion and without target lesion reintervention (TLR) within 1, 6 and 12 month
Freedom from SAE | Day 1, 1 month
  Freedom from SAE at discharge/30 days
All-cause mortality | 1 month, 6 months, 12 moths
  All-cause mortality at 1, 6 and 12 months;
Freedom from Clinically-driven TLR | 1 month, 6 months, 12 months
  Freedom from Clinically-driven TLR at 30 days, 6 and 12 months (any TLR for symptoms or ABI decrease > 30%; Clinically-driven Target Lesion Revascularization (CD-TLR) defined as any surgical or percutaneous intervention to the target lesion(s) after the index procedure
Rutherford shift | 1 month, 6 months, 12 months
  Rutherford shift from procedure at 30 days, 6 and 12 months (for AIOD subgroup)
Device Success | Day 1
  Device Success, defined as correct placement of the catheter and delivery of IVL (inflating balloon-delivering sonic pressure waves-deflating balloon) and recovery of the undamaged catheter;
Procedural Success | Day 1
  Procedural Success, defined as the presence of a residual stenosis < 50% (without stents and/or iliac limbs) or ≤ 30% (with stents and/or iliac limbs) by completion angiogram estimation;
Clinical Success | Day 1, 1 month
  Clinical Success, defined as procedural success without SAE before discharge
Freedom from procedure related complications | Day 1
  Freedom from procedure related complications
CASS score (exploratory endpoint) | Baseline
  Calcified Access Severity Score (CASS) at baseline CASS (Calcified Access Severity Score) multifactorial severity scale, which can be referred to for the definition of iliac access hostility

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Fazzini, MD, Principal Investigator — Fondazione PTV - Policlinico Tor Vergata; Pierluigi Antignani, MD, Study Chair — Fondazione Italiana Vascolare (FIV); Gabriele Morselli, PharmD, Study Director — EndoCore Lab
Locations (5):
- Italy (5):
  - Sant'Orsola Hospital, Bologna, Emilia-Romagna
  - Fondazione PTV - Policlinico Tor Vergata, Rome, Lazio
  - Ospedale San Giovanni di Dio, Florence, Tuscany
  - Ospedale Santa Maria della Misericordia di Perugia, Perugia, Umbria
  - Azienda Ospedaliero-Universitaria di Padova, Padua, Veneto